Study Title: Acceptance and Commitment Therapy for Tobacco Cessation Among Psychiatric Partial hospital Patients

NCT#: NCT03911960

Date: July 1st, 2020

Data analysis.

Due to small sample sizes, analyses will be descriptive.

- Aim 1. To assess the <u>feasibility</u> of the proposed ACT-based counseling program, we will conduct descriptive statistics on number of patients recruited to the program during the enrollment period compared to number of smokers in seen in the PHP during the enrollment period. In addition, we will conduct descriptive statistics on the number of sessions completed per group and rates of completion of the follow-up visit. To assess <u>acceptability</u> of the program, we will report descriptive statistics of responses on the Client Satisfaction Questionnaire in each group. To evaluate the <u>safety</u> of offering a tobacco cessation intervention during a PHP, we will report on the number of participants in the trial who are rehospitalized for a psychiatric reason during the treatment period based on participant self-report at end of treatment. To assess for symptom exacerbation we will report means of psychiatric symptoms by group pre and post intervention among those who completed follow-up.
- <u>Aim 2.</u> To evaluate for preliminary evidence of <u>efficacy</u>, we will report abstinence rates by group at end of treatment. Those lost to follow-up will be considered smokers.
- <u>Aim 3.</u> To assess for the effect of treatment condition on ACT treatment targets, we will report descriptive statistics of treatment targets before treatment and at follow-up for those who completed the follow-up visit.